CLINICAL TRIAL: NCT01310517
Title: Comparison of Very Low Contrast Volume Hand Injected Ventriculography to Standard Contrast Volume Power Injected Left Ventriculography From the Radial Artery Approach for Estimation of Left Ventricular Ejection Fraction.
Brief Title: Hand Injected Ventriculography vs. Power Injected Left Ventriculography
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to low enrollment.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Anthony Hilliard, Cardiology, Loma Linda University
Other Study IDs: HLVG2011
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Heart; Functional Disturbance
Keywords: Angiogram; Injected Contrast; Heart Function; contrast dye

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radial Coronary Angiography: The subjects enrolled in this study will be adults referred for radial coronary angiography with left ventriculography for clinical indications.

SUMMARY:
The purpose of the study is to directly compare two methods of evaluating heart function at the time of your angiogram. In both methods contrast dye is injected into the main heart chamber during the angiogram while x-ray images are taken. One method uses an automatic power injector to deliver the normal volume of contrast; the other method uses hand injection of very low volume of contrast into the main heart chamber. It is hypothesized that hand injection will prove to be an accurate method to estimate ejection fraction (EF) at the time of radial coronary angiography when compared directly to Power LV.

DETAILED DESCRIPTION:
Left ventriculography is a routine and accurate method of evaluating left ventricular ejection fraction (EF) at the time of coronary angiography. Power injected left ventriculography (Power LV) using standard volume (36 ml over 3 seconds) of contrast through a 5 Fr. angled pigtail catheter in the left ventricle is currently a routine clinical practice during left heart catheterization via the radial artery. With coronary angiography from the radial approach increasing in popularity there is a growing interest in hand injected left ventriculography (Hand LV) using a very low volume (8ml) of contrast through a 5 Fr. radial angiographic catheter. Potential benefits of this method include reduced contrast load, reduced procedure time and overall reduction in cost (less catheters used per procedure) as the procedure can be completed using a single diagnostic catheter. Potential limitations of this method include reduced opacification of the left ventricle and decreased number of cardiac cycles available to estimate EF. It is currently unknown if Hand LV is accurate in estimating EF when compared to the standard Power LV.

Objective: The primary objective of this study is to directly compare the accuracy of the very low volume Hand LV to the standard volume Power LV in estimating EF.

Methods: This study will be conducted in an outpatient setting. The subjects enrolled in this study will be adults referred for radial coronary angiography with left ventriculography for clinical indications. Subjects will undergo both Hand LV and Power LV at the time of angiography. EF for both Hand LV and Power LV will be estimated for each subject in a blinded fashion by 2 independent experienced cardiologists. Additionally, quantitative EF measurements will be made using integrated standard computer software for both the Power LV and the Hand LV. Each patient will serve as their own control.

Research Design: This is a prospective single center study designed to evaluate clinical techniques for diagnostic accuracy.

Clinical Relationships: It is anticipated that Hand LV will be and accurate method to estimate EF when compared to Power LV. (e.g. within a 5% difference is clinically is considered within inter and intra-individual variability.) This knowledge will allow clinicians to confidently perform Hand LV at the time of radial coronary angiography to estimate EF, reducing procedure time, contrast load and overall cost of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than 18 years of age referred for radial coronary angiography with left ventriculography for clinical indications at the Loma Linda Heart and Surgical Hospital or the Loma Linda University Medical Center will be included in this study.

Exclusion Criteria:

* Patients with a prosthetic aortic valve
* Patients with severe aortic stenosis
* Patients with suspected left main coronary artery disease
* Patients with other contraindications to left ventriculography.
* Patients with chronic kidney disease with a baseline creatinine ≥2.0 mg/dl if not already on renal replacement therapy will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects enrolled in this study will be adults referred for radial coronary angiography with left ventriculography for clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Imaging comparison | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Hilliard, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States